CLINICAL TRIAL: NCT03963479
Title: Vitamin B6 and Magnesium on Neurobehavioral Status of Autism Spectrum Disorder: A Randomized, Double-Blind, Placebo Controlled Study
Brief Title: Vitamin B6 and Magnesium- A Clinical Trial on ASD Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr. Farhana Khan, Resident, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: BSMMU/2018/14607
Record Dates: First submitted 2019-05-15; First posted 2019-05-24 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-05

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Magnesium; Vitamin B 6

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium-Vitamin B6 (Active Comparator): Magnesium (50mg) for ages 1-3 years (100mg) for ages 4-8 years (200mg) for ages 9-12 years Vitamin B6 (25mg) for ages 1-3 years (50mg) for ages 4-8 years (100mg) for ages 9-12years
  Interventions: Combination Product: Magnesium and Vitamin B6
- Placebo (Placebo Comparator): Magnesium (50mg) for ages 1-3 years (100mg) for ages 4-8 years (200mg) for ages 9-12 years Vitamin B6 (25mg) for ages 1-3 years (50mg) for ages 4-8 years (100mg) for ages 9-12years
  Interventions: Combination Product: Magnesium and Vitamin B6

INTERVENTIONS:
Combination Product: Magnesium and Vitamin B6 — Magnesium and Vitamin B6 will be given to the enrolled patients for 3 months

SUMMARY:
To determine whether Vitamin B6 and Magnesium improve neurobehavioral status in terms of General observation, Cognitive working, Socialization, Communication and Sensory Dysfunction in patient with Autism Spectrum Disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Children between 2 to 12 years of age suspected ASD assessed by DSM-5 and ADCL tool
2. Each patient will be free of psychoactive medication for atleast 3 months prior to the entry into the trial
3. Newly diagnosed patient
4. Co-morbid neurological disorder like hyperactivity

Exclusion Criteria:

1. Patients with chronic diseases or any known metabolic or hormonal diseases
2. Patients with any known chromosomal or genetic syndromes
3. Patients unable to give informed consent
4. Patients unable to travel to clinical visits or non co-operative

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
Autism Spectrum Disorder | 3 months
  General observation, Cognitive Working, socialization, Communication, Sensory Dysfunction.
  At first a autism will be diagnosed by DSM-5 .Then the above mention criterias along with the severity will be diagnosed by Autism Diagnostic Checklist tool by a psychologist.

SECONDARY OUTCOMES:
Autism Spectrum Disorder | 0 month
  The Autism Diagnostic Checklist will be repeated to compare the outcomes in terms of General observation, Cognitive Working, socialization, Communication, Sensory along with the severity of the Autism.

CONTACTS AND LOCATIONS:
Locations (1):
- Farhana Khan, Dhaka, Bangladesh